CLINICAL TRIAL: NCT02359422
Title: Randomized Control Trial Efficacy Study of a Comprehensive Sexual Health Media Literacy Education Program for Middle School Students
Brief Title: Evaluation of a Middle School Comprehensive Sexual Health Media Literacy Education Program
Acronym: MASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovation Research & Training (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: iRT-2R44HD061193-02-RCT; 2R44HD061193-02 (NIH)
Record Dates: First submitted 2014-09-03; First posted 2015-02-10 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Safe Sex
MeSH Terms: conditions — Safe Sex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Media Aware-Sexual Health (Experimental): 10-lesson middle school, comprehensive sexual health program developed based upon the Message Interpretation Processing model designed to increase critical thinking skills about media messages and reduce risky sexual behaviors.
  Interventions: Behavioral: Media Aware-Sexual Health
- Wait-list control (No Intervention)

INTERVENTIONS:
Behavioral: Media Aware-Sexual Health — 10-lesson middle school, comprehensive sexual health media literacy education program. Each lesson take approximately 50 minutes to teach and will be taught every school day for 2 weeks.
  Arms: Media Aware-Sexual Health

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial of a media literacy education program for middle school students with the goal of enhancing decision-making skills to prevent early and risky sexual behavior and teen pregnancy, and encourage healthy relationships.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to read and write in English

Exclusion Criteria:

* None

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1017 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in self-reported sexual activity assessed via questionnaire. | 2 weeks
Change in self-reported sexual activity assessed via questionnaire. | 3 months

SECONDARY OUTCOMES:
Change in self-reported intentions to engage in sexual activity assessed via questionnaire. | 2 weeks
Change in self-reported intentions to engage in sexual activity assessed via questionnaire. | 3 months
Change in self-reported attitude toward sexual activity assessed via questionnaire. | 2 weeks
Change in self-reported attitude toward sexual activity assessed via questionnaire. | 3 months
Change in self-reported attitudes toward contraception assessed via questionnaire. | 2 weeks
Change in self-reported attitudes toward contraception assessed via questionnaire. | 3 months
Change in self-reported attitude toward sexual communication assessed via questionnaire. | 2 weeks
Change in self-reported attitude toward sexual communication assessed via questionnaire. | 3 months
Change in self-reported perceived norms regarding sexual activity assessed via questionnaire. | 2 weeks
Change in self-reported perceived norms regarding sexual activity assessed via questionnaire. | 3 months
Change in self-reported perceived norms regarding contraception assessed via questionnaire. | 2 weeks
Change in self-reported perceived norms regarding contraception assessed via questionnaire. | 3 months
Change in self-reported perceived norms regarding sexual communication assessed via questionnaire. | 2 weeks
Change in self-reported perceived norms regarding sexual communication assessed via questionnaire. | 3 months
Change in self-reported self-efficacy to refusal sexual activity assessed via questionnaire. | 2 weeks
Change in self-reported self-efficacy to refusal sexual activity assessed via questionnaire. | 3 months
Change in self-reported self-efficacy to use contraception assessed via questionnaire. | 2 weeks
Change in self-reported self-efficacy to use contraception assessed via questionnaire. | 3 months
Change in self-reported self-efficacy for sexual communication assessed via questionnaire. | 2 weeks
Change in self-reported self-efficacy for sexual communication assessed via questionnaire. | 3 months
Change in self-reported intentions for condom/contraception use assessed via questionnaire. | 2 weeks
Change in self-reported intentions for condom/contraception use assessed via questionnaire. | 3 months
Change in self-reported intentions for sexual communication assessed via questionnaire. | 2 weeks
Change in self-reported intentions for sexual communication assessed via questionnaire. | 3 months

OTHER OUTCOMES:
Change in media deconstruction skills assessed via questionnaire. | 2 weeks
Change in media deconstruction skills assessed via questionnaire. | 3 months
Change in perceived realism of media messages assessed via questionnaire. | 2 weeks
Change in perceived realism of media messages assessed via questionnaire. | 3 months
Change in perceived similarity to media messages assessed via questionnaire. | 2 weeks
Change in perceived similarity to media messages assessed via questionnaire. | 3 months
Change in perceived desirability of media messages assessed via questionnaire. | 2 weeks
Change in perceived desirability of media messages assessed via questionnaire. | 3 months
Change in media skepticism assessed via self-report questionnaire. | 2 weeks
Change in media skepticism assessed via self-report questionnaire. | 3 months
Change in identification to media messages assessed via questionnaire. | 2 weeks
Change in identification to media messages assessed via questionnaire. | 3 months
Change in acceptance of dating violence norms assessed via questionnaire. | 2 weeks
Change in acceptance of dating violence norms assessed via questionnaire. | 3 months
Change in acceptance of gender role norms assessed via questionnaire. | 2 weeks
Change in acceptance of gender role norms assessed via questionnaire. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tracy M Scull, PhD, Principal Investigator — Innovation Research & Training
Locations (1):
- innovation Research & Training, Durham, North Carolina, United States

REFERENCES:
- [Derived] Scull TM, Kupersmidt JB, Malik CV, Morgan-Lopez AA. Using Media Literacy Education for Adolescent Sexual Health Promotion in Middle School: Randomized Control Trial of Media Aware. J Health Commun. 2018;23(12):1051-1063. doi: 10.1080/10810730.2018.1548669. Epub 2018 Nov 23. PMID 30468408